CLINICAL TRIAL: NCT01000077
Title: Establishment of Cell Culture Systems From Discarded Operating Room Tissue
Status: Enrolling by invitation | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB00007586
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Surgery
Keywords: Regenerative Medicine; Tissue Collection; Cell Culture Systems; Routine Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Healthy and diseased tissue will be harvested from tissue routinely discarded in the NCBH operating rooms, or from delivery rooms at Forsyth Medical Center during routine operative or childbirth procedures
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Discarded Operating Room Tissue: The purpose of this research study is to use the discarded (tissue that would normally be thrown out) tissue from your surgery in order to obtain cells that can be grown in a laboratory to study how to use cells like these to fix sick and diseased organs. We will test if these cells can be used to build new and healthy tissues. This technique is called tissue engineering. In this study we will be comparing cells obtained from different individuals.
- Discarded Placenta: During a standard surgery or delivery of a baby unneeded tissue is usually discarded. We would like to explore the opportunity to grow the cells of these discarded tissues in the laboratory. The cells will be placed in special dishes and supplemented with a mixture of salts and nutrients that were designed to allow the cells to survive outside the body and grow. This procedure is called tissue culture of cells. We will attempt to isolate a population of cells from the tissue culture and study them in the laboratory.

SUMMARY:
The purpose of this study is to establish viable cell culture system techniques for a variety of healthy and diseased tissues for use in future in vitro and in vivo research studies in tissue engineering.

DETAILED DESCRIPTION:
Healthy and diseased tissue will be harvested from tissue routinely discarded in the NCBH operating rooms, or from delivery rooms at Forsyth Medical Center during routine operative or childbirth procedures. Samples will be identified by source and disease state only. Disease state may be of several types including inflammation, malignancy, fibrosis, atherosclerosis, hyperplasia etc. These tissue samples will be promptly transported under sterile conditions to the Institute of Regenerative Medicine. The tissues will be broken down into individual cells by mechanical or enzymatic methods, diluted with growth media and inoculated onto sterile tissue culture flasks. The flasks will be placed into a 4% CO2 incubator for culture. The cultures will be cultivated for primary and progenitor cells and eventual RNA extraction and expression profiling. These cell lines may be then used for future in vitro and in vivo research studies yet to be determined. An Institutional Review Board (IRB) must approve any future research study using these tissue samples.

Source of Specimens:

Healthy and diseased tissue from a variety of sources (examples include bladder, foreskin, heart valves, blood vessels, prostate, kidney, uterus, ovary, salivary gland tissue, lacrimal gland tissue, muscle tissue, epithelial tissue, nerve tissue and vascular tissue from patients undergoing surgery) will be harvested from tissue routinely discarded in the NCBH operating rooms during routine operative procedures. In addition, normal term placentas will be obtained following vaginal deliveries at Forsyth Medical Center. No patient identifying information will be retained. No attempt will be made to match established cell lines derived from the tissue samples with the source patient. Eligibility for the protocol is restricted to an indication for surgical excision of the tissue in question.

Confidentiality Considerations:

No patient identifiers will be collected. It will not be possible to identify or link any tissue to the individual patient source in any way once it has been delivered to the Institute. The only information identifying the specimen will be tissue source, age and sex of patient, and disease state (if any). Informed consent will be obtained.

Sample Size:

Approximately 1000 people will take part in this study, all of them at Wake Forest University Health Sciences or Forsyth Medical Center.

ELIGIBILITY:
Eligibility Criteria:

* The subjects would include anyone undergoing a surgical procedure by one the of the surgeon co-investigators, during which discard tissue may be harvested.

Ages: 28 Days to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There is no specific study population for the this study. The patients from whom discarded tissue will be harvested will be any patients within the set age criteria in the operating room that have viable tissue excised for discard. In other words, when any investigators from the study have discard tissue as a result of a surgical procedure, this tissue will be a possible specimen for use in the protocol. Only discard tissue will be used, however, so if the tissue isn't used in the study, it would simply be thrown away.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-02 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steve J Hodges, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States